CLINICAL TRIAL: NCT03850873
Title: A Phase I Clinical， Tolerance and Pharmacokinetic Evaluation of 1 Schedules of Oral TQB3616，A Cyclin-Dependent Kinase Inhibitor ，In Patients With Advanced Breast Cancer
Brief Title: A Phase I Study of TQB3616 on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-I-0001
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3616 (Experimental): TQB3616 administerde days 28 of a 28-day schedule,doses ranging from 20m to 120mg once daily
  Interventions: Drug: TQB3616

INTERVENTIONS:
Drug: TQB3616 — TQB3616 administerde days 28 of a 28-day schedule,doses ranging from 20m，40mg，60mg，80mg，100mg，120mg once daily

SUMMARY:
TQB3616 may work in cancer by stopping cancer cells from multiplying.TQB3616 is in a new class of drugs called CDK inhibitors.This research study is the first time that TQB3616 will be given to people.TQB3616 is taken by mouth daily.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Patients definitely diagnosed by pathology and/or cytology as advanced breast cancer with ER+、Her2-,who failed with standard endocrine therapy.
3. ECOG PS:0-1,Survival is expected to be greater than 3 months
4. Main organs function is normal or must meet the following criteria(within past 14 days) 1) hemoglobin≥90g/L; neutrophils≥1.5 x109/L; Platelets≥100 x109/L 2)Albumin≥29g/L; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase(AST) and alanine transaminase(ALT)≤2.5 ULN, and ≤ 5 x ULN with hepatic metastasis;serum creatinine ≤1.5 xULN，creatinine clearance >60ml/min; Triglyceride≤3.0mmol/L, cholesterol≤7.75mmol/L

3)Doppler ultrasound evaluation: Left ventricular ejection fraction(LVEF)≥50% 5.Patients should be voluntary and sign the informed consent before taking part in the study

Exclusion Criteria:

1. Patients with malignant tumors, except for Cured cutaneous basal cell carcinoma and cervical carcinoma in situ
2. Prior treatment with chemotherapy with cytotoxic drugs within 4 weeks, mitomycin C or nirtosocarbamide within 8 weeks
3. Prior treatment with any anti-cancer therapy including hormone therapy radioimmunotherapy, molecular targeted therapy, immunotherapy or other biological therapy with 2 weeks
4. Patients treated with other CDK4/6 inhibitors;
5. Patients with brain metastasis, spinal cord compression, cancerous meningitis, CT or MRI examination reminds patients with cerebral or soft meningeal diseases in the screening phase;
6. Previous history of stem cell or bowe marrow transplant;
7. A variety of factors that affect oral medication (such as inability to swallow, gastrointestinal resection, intestinal obstruction, etc.)
8. Patients with non-healing wounds or fractures, except for bone metastatics with pathologic frature
9. Previous history of uncontrolled cardiovascular disease including: a) Grade 3 or higher congestive heart failure (NYHA Classification);b)unstable angina pectoris or newly developped angina pectoris within 3months before the trial; c) Myocardial in farction or stroke occured within 6 months prior to intiation of trial; d) Arrhythmias requiring antiarrhythmic treatment(beta-blocker or digoxin is permitted)
10. Patients who need to take CYP3A4 inhibitors or inducers from the screening period;
11. Patients with drug abuse history or unable to get rid of drugs or Patients with mental disorders
12. Patients with the urine protein≥2+, total ammount of 24 hours urinary protein determination>1.0 grams;
13. Patients with hyperactive/venous thrombosis events within 6 months,such as cerebrovascular accidents (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism
14. Patients with active hepatitis b or c infection
15. Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history;
16. Patients allergic to TQB3616 or any adjuvant in the capsule
17. Patients who took part in other trials within 4 weeks;
18. Patients with concomitant diseases which could seriously endanger themselves or those who won't complete the study according to investigators;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
DLT | Baseline up to 28 days
  Dose-Limiting Toxicities
MTD | Baseline up to 28 days
  Maximum Tolerated Dose

SECONDARY OUTCOMES:
Cmax | Hour 0(pre-dose),1,2,4,6,8,12,24,36,48,72,120,168hours post-dose on single dose ; Hour 0(pre-dose) of day1,day7,day14,day21,day28 on multiple dose and Hour 0(pre-dose),1,2,4,6,8,12,24hours post-dose on multiple dose of day28
  Maximum Observed Plasma Concentration
Tmax | Hour 0(pre-dose),1,2,4,6,8,12,24,36,48,72,120,168hours post-dose on single dose ; Hour 0(pre-dose) of day1,day7,day14,day21,day28 on multiple dose and Hour 0(pre-dose),1,2,4,6,8,12,24hours post-dose on multiple dose of day28
  Maximum Observed Plasma Concentration
t1/2 | Hour 0(pre-dose),1,2,4,6,8,12,24,36,48,72,120,168hours post-dose on single dose ; Hour 0(pre-dose) of day1,day7,day14,day21,day28 on multiple dose and Hour 0(pre-dose),1,2,4,6,8,12,24hours post-dose on multiple dose of day28
  Terminal Half-life
AUC | Hour 0(pre-dose),1,2,4,6,8,12,24,36,48,72,120,168hours post-dose on single dose ; Hour 0(pre-dose) of day1,day7,day14,day21,day28 on multiple dose and Hour 0(pre-dose),1,2,4,6,8,12,24hours post-dose on multiple dose of day28
  Area Under the Curve